CLINICAL TRIAL: NCT06100705
Title: A Single Arm Open-label, Phase II Study of Sipuleucel-T With Bipolar Androgen Therapy in Men With Metastatic Castration-resistant Prostate Cancer
Brief Title: Sipuleucel-T Combined With Bipolar Androgen Therapy in Men With mCRPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Dendreon (Industry)
Responsible Party: Principal Investigator, Joseph W Kim, Associate Professor of Internal Medicine (Medical Oncology), Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000035188
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Sipuleucel-T; Bipolar Androgen Therapy
MeSH Terms: interventions — testosterone 17 beta-cypionate; sipuleucel-T

STUDY DESIGN:
Intervention Model Description: open-label, single-arm phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Testosterone Cypionate + Sipuleucel-T (Experimental): Participants will start with testosterone injection every 4 weeks. The first dose of standard of care Sipuleucel-T will be prepared and infused after two doses of testosterone and will continue every 2 weeks for a total of 3 infusions at a standard schedule. The testosterone injection will continue once every 4 weeks until treatment discontinuation criteria are met.
  Interventions: Drug: Testosterone Cypionate; Drug: Sipuleucel-T

INTERVENTIONS:
Drug: Testosterone Cypionate — Testosterone Cypionate is an androgen and anabolic steroid medication which is used mainly in the treatment of low testosterone levels in men.
  Other Names: DEPO-Testosterone
Drug: Sipuleucel-T — Sipuleucel-T is the first FDA-approved immunotherapy in treatment of mCRPC. It is a therapeutic cancer vaccine composed of activated autologous dendritic cells loaded with an engineered fusion protein of prostatic acid phosphatase and granulocyte-macrophage colony-stimulating factor, PAP-GMCSF, also called PA2024. This cellular product is prepared in three steps: (1) leukapheresis to isolate CD54+ dendritic cells, (2) the cells and harvested and cultured with PA2024 ex vivo, and (3) re-infusion of the activated DC into the original patient. The preparation and administration of this autologous cellular product are done every 2 weeks for a total of three infusions and is designed to elicit an immune response to prostatic acid phosphatase.
  Other Names: Provenge

SUMMARY:
This is an open-label, single-arm phase II study of bipolar androgen therapy (BAT) given in addition with standard of care Sipuleucel-T to determine the interferon (IFN) gamma Enzyme-linked Immunospot (ELISPOT) response rate to PA2024 (an engineered fusion protein of prostatic acid phosphatase and granulocyte-macrophage colony-stimulating factor which the activated autologous dendritic cells in the Sipuleucel-T vaccine are loaded with) in patients with metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
The primary endpoint is the immune response to PA2024 as measured by ELISPOT by week 26. This immunological endpoint was chosen as the primary based on the data showing the Sipuleucel-T immune parameters correlating with overall survival from the pooled analysis phase III trials of Sipuleucel-T (Sheikh NA et al. Cancer Immunol Immunother 2013). Secondary endpoints include other immune parameters related to the Sipuleucel-T, including (1) APC cumulative activation (CD54 upregulation), (2) APC number and (3) total nucleated cells (TNC) count, which also have correlated with survival outcomes and clinical endpoints, and (4) T cell proliferation response to PA2024 and PAP, (5) ex vivo cytokine profile and (6) humoral response to PA2024 and PAP, clinical endpoints including: (7) PSA50 response rate (PSA50 RR), (8) objective response rate (ORR), (9) radiographic progression-free survival (rPFS), and (10) overall survival (OS), (11) safety and tolerability. We hypothesize that BAT potentiates the anti-tumor immune response and enhances clinical outcomes when given before and concurrently with Sipuleucel-T. Secondarily, we also hypothesize that the clinical activity of BAT will increase with concurrent Sipuleucel-T, as measured by PSA50 response rate and objective response rate compared to historical controls.

Participants will start with testosterone injection every 4 weeks. The first dose of standard of care Sipuleucel-T will be prepared and infused after two doses of testosterone and will continue every 2 weeks for a total of 3 infusions at a standard schedule. The testosterone injection will continue once every 4 weeks until treatment discontinuation criteria are met.

The participants will be assessed with HPE, and PSA every 4 weeks, and radiographic assessment per PCWG3 every 12 weeks. DEPO-Testosterone (testosterone cypionate) IM injection will continue until disease progression, unacceptable toxicity, or withdrawal of consent to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to the initiation of study procedures.
* Patients who meet the US FDA-approved indication for Sipuleucel-T: for asymptomatic or minimally symptomatic mCRPC at the discretion of the treating investigator.
* Histologically confirmed adenocarcinoma of the prostate.
* Metastatic disease as evidenced by soft tissue and/or bony metastases on baseline bone scan and/or computed tomography (CT) scan or Magnetic Resonance Image (MRI).
* Progressive castration-resistant prostate cancer (CRCP): Participants must have current or historical evidence of disease progression concomitant with surgical or medical castration and during immediate past systemic therapy, as demonstrated by (a) PSA progression, or (b) progression of measurable disease, or (c) progression of non-measurable disease as defined below:

  1. By PSA: two consecutively rising PSA values, at least 7 days apart, each ≥ 1.0 ng/mL and ≥ 50% above the minimum PSA observed during castration therapy or above the pre-treatment value if there was no response.
  2. By measurable disease: Progressive disease by RECIST v1.1 criteria
  3. By non-measurable disease

  i. Soft tissue disease: The appearance of 1 or more new lesions, and/or unequivocal worsening of non-measurable disease when compared to imaging studies acquired during castration therapy or against the pre-castration studies if there was no response.

ii. Bone disease: Appearance of 2 or more new areas of abnormal uptake on bone scan when compared to imaging studies acquired during castration therapy or against the pre-castration studies if there was no response. Increased uptake of pre-existing lesions on bone scan does not constitute progression.

* Castration status confirmed by serum testosterone level <50ng/dL
* ECOG Performance Status of 0 or 1.
* Adequate liver function:

  1. Bilirubin <2.0 x institutional upper limit of normal (UNL)
  2. AST (SGOT) <2.5 x UNL
  3. ALT (SGPT) <2.5 x UNL
* Acceptable renal function

  a) Serum creatinine <2.0 x UNL
* Acceptable hematologic function:

  1. Absolute neutrophil count (ANC) > 1.0 x10^9 cells /L)
  2. Platelet counts > 100 x 10^9 / L)
  3. Hemoglobin >9 g/dL

Exclusion Criteria:

* PSA >20ng/dL within the 4 weeks prior to signing ICF
* Previously treated with three or more FDA-approved androgen/AR signaling inhibitors (ASI) (e.g., abiraterone, enzalutamide, apalutamide, darolutamide). No minimum number of ASI is required.
* Prior chemotherapy for mCRPC. However, prior chemotherapy administered for mCSPC is allowed unless the disease progression to CRPC occurred within 12 months from the last dose of chemotherapy.
* Prior treatment with Sipuleucel-T or supraphysiologic dose of testosterone treatment for prostate cancer.
* Prior systemic treatment with ASI, PARP inhibitor or Radium-223 or other systemic anti-cancer therapy for prostate cancer within 4 weeks prior to start of treatment.
* Prior prednisone >10mg (or its equivalent) within 2 weeks prior to registration.
* Prior immunotherapy or Lu177 PSMA radioligand therapy within 6 weeks prior to registration.
* Prior palliative radiotherapy within 2 weeks prior to registration.
* Radiographic evidence of hepatic metastases
* Use of narcotics including tramadol or stronger for cancer-related pain within 4 weeks prior to signing ICF. Use of NSAIDs or acetaminophen is allowed.
* Active autoimmune disease requiring systemic corticosteroids of prednisone greater than 10mg a day or the equivalent dose of other corticosteroids.
* Known active HIV, Hepatitis B or Hepatitis C or Human T cell Lymphotropic virus (HTLV)-1 infection. Testing is not required. Note: Participants with resolved, historic HIV, Hepatitis B or Hepatitis C or Human T cell Lymphotropic virus (HTLV)-1 will be assessed by the PI and deemed eligible if their viral infections are in remission: without detectable viruses and secondary immunodeficiency, and without requiring any treatments that affects immune function. Eligibility will be determined after a discussion with the PI and adequate standard clinical tests are acquired to prove that they are in remission.
* Active infection requiring parenteral antibiotic therapy or causing fever (temperature >100.5 in Fahrenheit scale) within 1 week prior to registration.
* Life expectancy of less than 6 months prior to signing ICF.
* Any medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence with study requirements or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To determine the immune response to PA2024 with BAT and Sipuleucel-T | Through the study completion, average 12 months
  As measured by ELISPOT from blood samples in pg/ml

SECONDARY OUTCOMES:
To determine antigen presenting cell (APC) cumulative activation | Through the study completion, average 12 months
  as assessed by flow cytometry staining and defined as the increase in surface CD54 on APCs, expressed as an upregulation ratio of the average number of molecules on after culture versus before culture cells from the sipuleucel-T product from blood samples in pg/ml
To determine APC number | Through the study completion, average 12 months
  as assessed by flow cytometry staining from each sipuleucel-T product. from blood samples in pg/ml
To determine total nucleated cell count | Through the study completion, average 12 months
  as assessed by flow cytometry staining from each sipuleucel-T product. from blood samples in pg/ml
To determine T cell proliferation to PA2024 | Through the study completion, average 12 months
  As measured by ELISPOT from blood samples in pg/ml
To determine T cell proliferation to Prostatic Acid Phosphatase (PAP) | Through the study completion, average 12 months
  As assessed by tritiated thymidine uptake from blood samples
To determine ex vivo cytokine profiles with BAT + Sipuleucel-T | Through the study completion, average 12 months
  As assessed via Luminex assay from blood samples in pg/ml
To determine humeral response with BAT + Sipuleucel-T | Through the study completion, average 12 months
  As assessed by ELISA from blood samples in pg/ml
To determine PSA50 response rate to BAT + Sipuleucel-T | Through the study completion, average 12 months
  As defined by PSA decline > 50% from baseline at any point
To determine objective response rate (ORR) to BAT + Sipuleucel-T | Through the study completion, average 12 months
  As defined by RECIST v1.1 criteria
To estimate radiographic progression free survival (rPFS) | From the date of registration until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 5 years
  Defined as the time interval from registration to the first occurrence of radiographic progression by Tc99 Bone Scan using PCWG3 criteria or radiographic soft tissue progression by RECIST v1.1 or death from any cause, whichever occurs first.
To estimate overall survival (OS) | From the date of registration until the date of death from any cause, assessed up to 5 years
  Defined as the time interval from registration to death due to any cause
To assess safety and tolerability to BAT+ Sipuleucel-T | Through the study completion, average 12 months
  As assessed by using CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Kim, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States